CLINICAL TRIAL: NCT02363556
Title: A Factorial-Design Randomized Controlled Trial Comparing Misoprostol Alone to Dilapan With Misoprostol and Comparing Buccal to Vaginal Misoprostol for Same-Day Cervical Preparation Prior to Dilation & Evacuation
Brief Title: Comparing Misoprostol Alone to Dilapan With Misoprostol and Comparing Buccal to Vaginal Misoprostol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Matthew Reeves, MD, Medstar Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2014-110
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Second Trimester Abortions
Keywords: Cervical Dilation; Dilation and Evacuation; Misoprostol; Misoprostol-Dilapan; Abortion
MeSH Terms: conditions — Dilatation, Pathologic | interventions — dilapan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol Alone (Experimental): Subjects enrolled into this arm of the study will receive misoprostol 400-mcg only.
  Interventions: Procedure: Misoprostol administered vaginally; Procedure: Misoprostol administered buccally
- Dilapan with Misoprostol (Experimental): Subjects enrolled into this arm of the study will receive Dilapan with 400-mcg misoprostol.
  Interventions: Procedure: Misoprostol administered vaginally with Dilapan; Procedure: Misoprostol administered buccally with Dilapan

INTERVENTIONS:
Procedure: Misoprostol administered vaginally
  Arms: Misoprostol Alone
Procedure: Misoprostol administered buccally
  Arms: Misoprostol Alone
Procedure: Misoprostol administered vaginally with Dilapan
  Arms: Dilapan with Misoprostol
Procedure: Misoprostol administered buccally with Dilapan
  Arms: Dilapan with Misoprostol

SUMMARY:
This randomized controlled trial will use a 2 by 2 factorial design to assess methods of cervical preparation prior to Dilation and Evacuations (D&Es) at 14 0/7 to 19 6/7 weeks gestational age. In total, 160 woman will be randomized to misoprostol alone or Dilapan with misoprostol and separately randomized to buccal or vaginal administration of 400-mcg misoprostol. A total of 80 women will receive 400-mcg misoprostol only (40 vaginal and 40 buccal). Another 80 women will have Dilapan inserted and then use misoprostol (40 vaginal and 40 buccal). Four to six hours later, the Dilation and Evacuation (D&E) procedure will be performed.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the efficacy of same-day 400-mcg misoprostol alone to same-day Dilapan with 400-mcg misoprostol for cervical preparation prior to D&E at 14 0/7 to 19 6/7 weeks. Patients will first be randomized to misoprostol alone or misoprostol-Dilapan, and then separately randomized to use the misoprostol buccally or vaginally.

The primary outcome measure is total procedure time. Secondary outcomes include D&E procedure time, initial cervical dilation (measured by the largest Hegar dilator accepted without resistance prior to the start of the procedure), patient-oriented outcomes (side effects of buccal and vaginal misoprostol), and patient acceptability and satisfaction.

The investigators have chosen a randomized controlled trial with a factorial design to be conducted at Washington Hospital Center and Planned Parenthood of Metropolitan Washington. A total up to 180 English speaking women will be enrolled in the study so that 160 will be randomized and receive study interventions. The study will enroll healthy women, over the age of 18, eligible for non-urgent D&E at 14 0/7 weeks to 19 6/7 weeks, confirmed by sonogram. The women will be randomized to receive either misoprostol alone or Dilapan with misoprostol. Women will then be randomized to receive 400-mcg of misoprostol either buccally or vaginally. Computer generated randomization will be utilized to assign treatment arms. Approximately 4-6 hours prior to procedure, women will be randomly assigned to one of the following treatment combinations:

1. Misoprostol 400-mcg vaginally
2. Misoprostol 400-mcg buccally
3. Dilapan insertion with 400-mcg misoprostol vaginally
4. Dilapan insertion with 400-mcg misoprostol buccally

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* 18 years of age or older
* Eligible for non-urgent Dilation and Evacuations at 14 0/7 - 19 6/7 weeks gestation confirmed by sonogram.

Exclusion Criteria:

* Women who do not speak English.
* Fetal demise
* Intolerance, allergy or contraindication to misoprostol or Dilapan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Total procedure time | 4-6hrs
  Total procedure time is defined as the time required for dilator insertion plus the D&E time.

SECONDARY OUTCOMES:
D&E procedure time | 0-60 mins
Initial cervical dilation | 0-10 mins
  Measured by the largest Hegar dilator accepted without resistance prior to the start of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Matthew Reeves, MD MPH, Principal Investigator — MedStar Washington Hospital Center & Planned Parenthood of Metropolitan Washington; Dr. Jamilah Shakir, MD MPH, Study Chair — Medstar Health Research Institute
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Planned Parenthood Metropolitan Washington, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No